CLINICAL TRIAL: NCT03541616
Title: Prevalence of Subclinical Atrial Fibrillation in High Risk Heart Failure Patients and Its Temporal Relationship With Hospital Readmission for Heart Failure
Brief Title: Prevalence of Subclinical Atrial Fibrillation in Heart Failure Patients and Its Relationship With Hospital Readmission
Acronym: PROTECT-HF
Status: Completed | Type: Observational
Sponsor: Population Health Research Institute (Other)
Collaborators: Heart and Stroke Foundation of Canada (Other); Canadian Cardiovascular Society (Other)
Responsible Party: Sponsor
Other Study IDs: PROTECT-HF
Record Dates: First submitted 2018-05-17; First posted 2018-05-30 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Heart Failure; Atrial Fibrillation
MeSH Terms: conditions — Heart Failure; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Enrolled Patients
  Interventions: Device: ECG Patch, pocket ECG monitor

INTERVENTIONS:
Device: ECG Patch, pocket ECG monitor — Two consecutive 14-day ECG monitor patches or one single 28-day pocket ECG monitor (28-days total monitoring) implemented at the time of hospital discharge .

SUMMARY:
Multicentre, prospective cohort study in patients with a history of HF with preserved or reduced ejection fraction admitted to hospital with acutely decompensated HF. Eligible and consenting patients will be enrolled at 3 Hamilton, Ontario area hospitals and receive 28-day ECG monitoring implemented at the time of hospital discharge. Patients will be followed for a total of 1 year from hospital discharge.

DETAILED DESCRIPTION:
In patients discharged from hospital after an admission for acute heart failure (HF) decompensation, subclinical atrial fibrillation (AF) of 30 minutes or greater in duration is common (at least 15% of patients without prior AF) and is associated with increased risk of re-hospitalization within 30-days.

Study Objectives:

1. To evaluate the prevalence of subclinical AF ≥30 minutes in duration in patients discharged from hospital following an admission for acute HF exacerbation and who have no known history of clinical AF.
2. To examine the temporal association between subclinical AF ≥30 minutes in duration and 30-day hospital readmission for HF.

ELIGIBILITY:
Inclusion Criteria:

1. Hospitalized with a most responsible diagnosis of acute decompensated heart failure.
2. Clinical signs and symptoms of heart failure as per the Boston criteria (i.e. score ≥8)

Exclusion Criteria:

1. History of clinical atrial fibrillation
2. History of hypertrophic cardiomyopathy or congenital heart disease.
3. End stage renal disease or advanced renal dysfunction (e.g. estimated glomerular filtration rate, eGFR < 15 mL/min/1.73 m2)
4. Cardiothoracic surgery in the past 30 days or imminently planned (does not include percutaneous procedures).
5. Unable or unwilling to provide informed consent.
6. Presence of a pacemaker or an ICD with an atrial lead (which can already diagnose AF).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a history of HF who are admitted to hospital with acutely decompensated HF and have no prior history of AF.
Sampling Method: Non-Probability Sample
Enrollment: 242 (Actual)
Dates: Start 2018-03-24 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2023-03-27 (Actual)

PRIMARY OUTCOMES:
Subclinical atrial fibrillation ≥30 minutes in duration | 30 days post-discharge

SECONDARY OUTCOMES:
Heart failure re-hospitalization | 30 days post-discharge

OTHER OUTCOMES:
Subclinical atrial fibrillation >6 minutes in duration | 30 days post-discharge
Clinical atrial fibrillation | 30 days post-discharge
Heart Failure re-hospitalization | 1 year post-discharge
All-cause re-hospitalization | 30 days and 1 year post-discharge
All-cause and cardiovascular mortality | 30 days and 1 year post-discharge
Incident stroke/TIA or systemic thromboembolism | 30 days and 1 year post-discharge
Myocardial infarction | 30 days and 1 year post-discharge
Patient acceptance of device monitoring | 30 days post-discharge
  Measured by simple questionnaire that has not been validated. Patients will be asked to respond to satisfaction questions on a scale of a) strongly agree b) agree c) somewhat agree d) disagree or e) strongly disagree. The questions will ask about their experience with the device, such as: were instructions on using the device clear, the device was easy to use, the device did not limit my usual daily activities, the size of the device was not cumbersome, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge A Wong, MD, MPH, Principal Investigator — Population Health Research Institute; Stuart Connolly, MD, Principal Investigator — Population Health Research Institute
Locations (5):
- Canada (5):
  - Hamilton General Hospital, Hamilton, Ontario
  - Juravinski Hospital, Hamilton, Ontario
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - St. Mary's Hospital, Kitchener, Ontario
  - St. Catherines General Hospital, St. Catharines, Ontario

IPD SHARING:
Plan to Share IPD: No